CLINICAL TRIAL: NCT02159794
Title: HLT transfemOral Replacement of aortIc Valve Via transcatherteriZatiON CANADA
Acronym: HORIZON CANADA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: HLT determined that design changes are necessary before reopening a study
Sponsor: HLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLT1401
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Severe Aortic Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Aortic valve stenosis; Severe aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HLT Transcatheter Aortic Valve System (Experimental): Transcatheter aortic valve replacement with an HLT Transcatheter Aortic Valve System
  Interventions: Device: HLT Transcatheter Aortic Valve System

INTERVENTIONS:
Device: HLT Transcatheter Aortic Valve System — Transcatheter aortic valve replacement with an HLT Transcatheter Aortic Valve System

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the HLT System in patients with severe aortic stenosis who present at High Risk for aortic valve replacement surgery.

DETAILED DESCRIPTION:
Prospective, non-randomized, single arm, single-center first-in-man feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

1. 75 years of age or older
2. Echocardiographic or hemodynamic based evidence of calcific (senile) aortic stenosis with one of the following: aortic valve EOA <1.0 cm2 or 0.6 cm2/m2 , mean aortic valve gradient >40 mmHg or peak aortic valve velocity >4 m/sec
3. Symptomatology due to aortic stenosis resulting in a New York Heart Association (NYHA) Functional Classification of II or greater
4. Aortic valve annular diameter ≥ 21 and ≤23mm measured by MSCT
5. An STS score ≥10; or Logistic EuroScore I ≥ 15; or a determination by one cardiovascular surgeon and one cardiologist that the co-morbidities not captured by the STS or EuroScore expected to increase the operative mortality risk to > 15%.
6. Geographically available, willing to comply with follow up and able to provide written informed consent

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve, or noncalcified aortic valve; or valve eccentricity (calcific or otherwise) that in the opinion of the investigator could compromise procedural success.
2. Pre-existing prosthetic heart valve in any position, or prosthetic ring
3. Severe (Grade 3 to 4) aortic, mitral or tricuspid valve regurgitation
4. Moderate to severe mitral stenosis
5. Myocardial infarction within the past 30 days*
6. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
7. LVEF < 30%
8. Uncontrolled hypertension (i.e. blood pressure at baseline > 140 mmHg systolic ; or in the opinion of the investigator cannot be controlled by medical therapy).
9. Severe pulmonary hypertension with pulmonary systolic pressure greater than two-thirds of systemic pressure
10. Hemodynamic instability requiring inotropic drug therapy within the past 14 days or mechanical support within the past 6 months*
11. Untreated clinically significant coronary artery disease requiring revascularization
12. Presence of significant aortic disease such as atheroma, thrombus, or aneurysm which, in the opinion of the investigator, precludes safe implant delivery
13. Blood dyscrasias defined as: acute leukopenia, acute anemia, acute thrombocytopenia, history of bleeding diathesis or coagulopathy
14. Patient ineligible for or refuses blood transfusions
15. Unfavorable peripheral vascular anatomy or disease (e.g. severe obstructive calcification, severe tortuosity or small vessels) that would preclude passage of catheters from the femoral arterial access to the aorta as evidenced by peripheral MSCT
16. Active peptic ulcer or gastrointestinal bleeding within the past 90 days*
17. Stroke or transient ischemic attack within past 6 months*
18. Renal insufficiency as demonstrated by a serum creatinine > 2.5 mg/dL or end stage renal disease requiring chronic dialysis
19. Active infection requiring ongoing treatment
20. Need for emergent surgery or intervention other than the investigational procedure
21. Any therapeutic invasive cardiac procedure performed or planned to perform within 30 days of the index procedure, (or 6 months for drug eluting coronary stent or biventricular pacemaker implantation)*
22. Hypersensitivity or contraindication to procedural medication and device materials (e.g. titanium, nickel, pork) which cannot be adequately pre-medicated
23. Life expectancy < 1 year due to non-cardiac co-morbid conditions
24. Currently participating in any investigational drug or device studies that may confound the results of this study
25. History of any cognitive or mental health status that would interfere with study participation * At the time of procedure, if a subject's medical status has changed since enrollment, the subject shall be re-evaluated for eligibility

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Procedural Device Performance | Post procedure (day of procedure)
  The primary performance endpoint is the Device Success defined as:
  * Absence of procedural mortality AND
  * Correct positioning of a single HLT Valve into the proper anatomical location AND
  * Intended performance of the HLT Valve (no prosthesis- patient mismatch and mean aortic valve gradient < 20 mmHg or peak aortic valve velocity < 3 m/sec, AND no moderate or severe aortic valve regurgitation)
Mortality | 30 days
  The primary safety objective is all-cause mortality at 30 days.

SECONDARY OUTCOMES:
Post-procedural Valve Performance | post procedure (day of procedure), pre-discharge (up to 14 days), 1, 6, 12, 24, 36, 48 and 60 months
  The HLT Valve performance will be evaluated by the following parameters with echocardiograms obtained at baseline, procedural, pre-discharge, 1, 6, 12, 24, 36, 48 and 60 months:
  * Aortic valve effective orifice area (EOA)
  * Severity of aortic valve regurgitation (AR)
  * Aortic valve gradient
Adverse Events | 5 years
  All adverse events will be assessed throughout the 5 year follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodés-Cabau, M.D., Principal Investigator — Quebec Heart and Lung Institute
Locations (1):
- Quebec Heart and Lung Institute, Québec, Quebec, Canada